CLINICAL TRIAL: NCT06678308
Title: Comparison of the Efficacy and Safety of Glue with Calibrated Microparticles in Prostatic Artery Embolisation As a Treatment for Symptomatic Benign Prostatic Hyperplasia.
Brief Title: Comparison of Glue with Microparticles in Prostatic Artery Embolization
Acronym: EMBOLICOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Almaviva Sante (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-08; ID-RCB number: 2024-A01753-44 (Other: ANSM)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magic Glue® (Experimental): Embolisation of the prostatic arteries will be performed with Magic Glue® combined with lipiodol
  Interventions: Device: Embolisation with Magic Glue®
- Embosphere® (Active Comparator): Embolisation of prostatic arteries will be performed with 300-500 micron trisacryl particles (Embosphere®)
  Interventions: Device: Embolisation with Embosphere®

INTERVENTIONS:
Device: Embolisation with Magic Glue® — Magic Glue® will be injected within prostatic arteries, leading to ischaemia and necrosis of part of the adenomatous tissue of the prostate gland
  Arms: Magic Glue®
Device: Embolisation with Embosphere® — Embosphere® will be injected within prostatic arteries, leading to ischaemia and necrosis of part of the adenomatous tissue of the prostate gland
  Arms: Embosphere®

SUMMARY:
Prostatic artery embolisation (PAE) is an alternative treatment to surgery for benign prostatic hyperplasia (BPH). It has been practised since 2012 and numerous publications have proved not only its safety but also its efficacy.

The principle of PAE is to occlude the prostatic arteries with an 'embolising agent', which will result in ischaemia and necrosis of part of the adenomatous tissue of the prostate.

The reference embolisation agent is a suspension of calibrated trisacryl microparticles 300-500 microns in size.

Recently, the use of glue has been retrospectively studied with acceptable efficacy and safety.

In this context, where only the results of retrospective studies are available, it is necessary to initiate comparative prospective studies to assess the efficacy and safety of the glue compared with calibrated microparticles.

DETAILED DESCRIPTION:
Prostatic artery embolisation (PAE) is an alternative treatment to surgery for benign prostatic hyperplasia (BPH), and its place is recognised in the recommendations of the Male Voiding Disorders Committee (French Urological Association). It has been practised since 2012 (Carnevale et al, 2020), and numerous publications have proved not only its safety but also its efficacy (Malling et al, 2019).

The principle of PAE is to occlude the prostatic arteries with an 'embolising agent', which will result in ischaemia and necrosis of part of the adenomatous tissue of the prostate.

The reference embolisation agent, used by the majority of expert prostate embolisation teams, is a suspension of calibrated trisacryl microparticles 300-500 microns in size.

Recently, the use of glue has been retrospectively studied with acceptable efficacy and safety (Loffroy et al, 2021). Another retrospective comparative study (Salet et al, 2022) reported no significant difference in clinical efficacy between the use of glue and 300-500 micron trisacryl particles.

In this context, where only the results of retrospective studies are available, it is necessary to initiate comparative prospective studies to assess the efficacy and safety of the glue compared with calibrated microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged ≥ 50 years and ≤ 80 years
* Patient with symptomatic BPH (prostatic volume ≥ 40 ml measured on prostatic MRI, IPSS ≥ 8, uroflowmetry < 15 ml/s).
* Patient failing or intolerant to drug treatment (tadalafil and/or one of the alpha-blockers, alfuzosin, tamsulosin, silodosin or doxazosin).

Exclusion Criteria:

* Patient with advanced and complicated BPH on renal and bladder ultrasound:

Severe obstruction related bladder wall lesions : >3 micro-diverticula or single or multiple diverticula with a sac diameter > 10 mm.

Chronic dilatation of the excretory cavities : diameter of one or both pyelons >15 mm.

* Patient with suspected prostate or bladder cancer on MRI
* Patients with moderate or severe chronic renal failure, with creatinine clearance < 40 ml/min.
* Patient with prostate or bladder cancer diagnosed by biopsy in the 6 months preceding the inclusion visit.
* Patient with an active urinary tract infection
* Patient already included and participating in another clinical study.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of embolisation | Month 3
  Efficacy of embolisation will be assessed with IPSS score (International Prostate Symptoms Score). IPSS questionnaire consists of 7 questions (ranging from 0 to 5) on mictional difficulties for a maximum total of 35 points (0 means no mictional difficulty).

SECONDARY OUTCOMES:
Post-Mictional Residue | Month 1, Month 3 and Month 12
  Post-Mictional Residue will be assessed will be measured in ml by ultrasound
Prostatic infarct areas | Month 3
  Prostatic infarct areas will be measured in mm3 on MRI
Sexual function | Month 1, Month 3 and Month 12
  Sexual function will be assessed with IIEF5 questionnaire (International Index of Erectile Function form 5) (0 - 25 points). Score lower than 10 means severe erectile dysfunction whereas score higher than 20 means normal erectile function.
Patient quality of life | Month 1, Month 3 and Month 12
  Patient quality of life will be assessed with IPSS quality of life question (1 - 7). 1 means patient is very satisfied of his/her quality of life
Prostatic Serum Antigen | Month 1, Month 3 and Month 12
  Prostatic Serum Antigen (PSA) will be measured from blood sample. Normal value should be lower than 4 ng/ml
Urinary flow | Month 1, Month 3 and Month 12
  Urinary flow will be measured in ml/s by flow measurement
Prostatic volume | Month 3 and Month 12
  Prostatic volume will be in ml on MRI
Efficacy of embolisation | Month 1 and Month 12
  Efficacy of embolisation will be assessed with IPSS score (International Prostate Symptoms Score). IPSS questionnaire consists of 7 questions (ranging from 0 to 5) on mictional difficulties for a maximum total of 35 points (0 means no mictional difficulty).
Safety of embolisation | Day 15, Month 3 and Month 12
  Safety of embolisation will be assessed with post-empbolisation symptoms description and other adverse events description

CONTACTS AND LOCATIONS:
Overall Officials: Grégory AMOUYAL, MD, Principal Investigator — Clinique de l'Alma
Locations (1):
- Clinique de l'Alma, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No